CLINICAL TRIAL: NCT01307592
Title: Pilot Study of GC. (Gemcitabine-Rituximab-Oxaliplatin Combination) Given Every 14 Days With Maintenance Lenalidomide for the Treatment of Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Gemcitabine Hydrochloride, Rituximab, Oxaliplatin, and Lenalidomide in Treating Patients With Relapsed or Refractory, Aggressive Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000695874; CAM-09-01; CELGENE-RV-NHL-PI-0452
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2011-02

CONDITIONS: Lymphoma
Keywords: peripheral T-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Gemcitabine; Lenalidomide; Oxaliplatin

INTERVENTIONS:
Biological: rituximab
Drug: gemcitabine hydrochloride
Drug: lenalidomide
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride, oxaliplatin, and , work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Lenalidomide may stop the growth of non-Hodgkin lymphoma by blocking blood flow to the cancer. Giving rituximab and chemotherapy together with lenalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab, gemcitabine hydrochloride, and oxaliplatin together with lenalidomide works in treating patients with relapsed or refractory, aggressive non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the rate of conversion to complete response (CR) after switching to lenalidomide in patients with relapsed or refractory, aggressive non-Hodgkin lymphoma whose maximum response to gemcitabine hydrochloride, rituximab, and oxaliplatin is a partial response (PR).

Secondary

* To determine the overall survival of these patients treated with this regimen.
* To determine the progression-free survival of patients with CR and PR.
* To determine the treatment-related toxicity of this regimen combination in these patients.

OUTLINE: This is a multicenter study.

* Rituximab, gemcitabine hydrochloride, and oxaliplatin: Patients with B-cell lymphoma receive rituximab IV on day 1; all patients receive gemcitabine hydrochloride IV over 30 minutes and oxaliplatin IV over 2 hours on day 1 or day 2*. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients with T-cell lymphoma proceed to chemotherapy on day 1 without receiving rituximab; patients with B-cell lymphoma receive chemotherapy on day 2.

Patients are reevaluated after 4 courses of therapy. Patients who achieve a complete response (CR) receive 2 more courses of therapy and then proceed to bone marrow transplantation (BMT); those that do not receive a BMT receive maintenance lenalidomide for 2 years. Patients who achieve a partial response (PR) and who are not candidate for autologous stem cell transplantation (ACT) are treated with lenalidomide**. Once patients with PR achieve a CR or < CR with lenalidomide treatment, they proceed to maintenance lenalidomide for 2 years, unless they become candidates for ACT***. Patients with stable disease or progressive disease after 4 courses of therapy are treated with lenalidomide, unless they become eligible for ACT***.

NOTE: **Patients in whom a delay of > 4 months would occur for ACT are treated with lenalidomide until 3 weeks prior to ACT.

NOTE: **Once eligible, patients proceed to ACT as soon as feasible.

* Maintenance lenalidomide: Patients receive oral lenalidomide once daily on days 1-21. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically for toxicity analysis.

After completion of study treatment, patients are followed up at 28 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed aggressive non-Hodgkin lymphoma, including any of the following subtypes:

  * Follicular large cell lymphoma
  * Diffuse large cell lymphoma
  * Peripheral T-cell lymphoma
  * Transformed lymphoma
  * Lymphoblastic lymphoma
  * Burkitt or Burkitt-like lymphoma
* Refractory or relapsed disease meeting the following criteria:

  * Patients who either did not respond to prior therapy or whose best response was partial response after ≥ 4 courses of chemotherapy
  * Histologic confirmation of relapsed or refractory disease is desirable but not mandatory and will be left to the discretion of the investigator
* Must have evaluable or measurable disease
* Patients who are candidates for stem cell or bone marrow transplantation allowed
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Absolute neutrophil count ≥ 1,000/mm³ (unless due to marrow infiltration by lymphoma)
* Platelet count ≥ 100,000/mm³ (unless thrombocytopenia is due to marrow infiltration by lymphoma)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) (unless liver is involved with lymphoma, hemolysis, or Gilbert syndrome)
* Serum creatinine ≤ 2.0 mg/dl or creatinine clearance ≥ 30 ml/min (unless creatinine elevation is due to lymphoma)
* ALT ≤ 2 times ULN (≤ 5 times ULN if liver metastasis is involved with lymphoma)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception for ≥ 28 days before, during, and for ≥ 28 days after completion of study therapy

  * Men must use latex condoms even after a successful vasectomy
* Must be enrolled in the mandatory RevAssist® program and be willing to comply with its requirements
* No neurosensory or neuromotor dysfunction ≥ grade 3
* No known HIV positivity or active hepatitis B or C (hepatitis B surface antigen positivity or hepatitis C RNA positivity)
* No known hypersensitivity to thalidomide or erythema nodosum characterized by desquamating rash while taking thalidomide or other similar drugs
* No history of allergy to platinum or any of its derivatives or E. coli-derived products
* No other malignancies within the past 5 years, except treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or any surgically cured malignancy from which the patient has been disease-free for ≥ 5 years
* No NYHA class III-IV congestive heat failure (no symptoms on less than ordinary exertion or at rest)
* No uncontrolled or intercurrent disease, including any of the following:

  * Arrhythmias
  * Angina pectoris
  * Active infection or fever > 38.2 C (unless due to lymphoma)
* No serious medical condition, laboratory abnormality, or psychiatric illness that would place patient at risk in study or confound ability to interpret study data

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior gemcitabine hydrochloride, oxaliplatin, or lenalidomide
* Prior rituximab allowed
* No more than 4 prior regimens of chemotherapy allowed, including stem cell or bone marrow transplantation
* More than 2 weeks since prior and no concurrent anticancer therapy, including radiotherapy, hormonal therapy, or surgery
* More than 3 weeks since prior chemotherapy or radiotherapy
* More than 28 days since prior and no other concurrent investigational drug trial or investigational agent
* Able to take aspirin (81 mg or 325 mg) daily or low molecular weight heparin as prophylactic anticoagulation
* No concurrent thalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion to complete response (CR) after switching to lenalidomide

SECONDARY OUTCOMES:
Overall survival
Progression-free survival
Safety of this regimen combination
Rate of conversion to partial response and CR of non-responders treated with lenalidomide

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — Auxilio Mutuo Cancer Center
Locations (1):
- Centro de Cancer del Hospital Auxilio Mutuo, San Juan, Puerto Rico